CLINICAL TRIAL: NCT07338799
Title: Effectiveness of Multimodal Therapy Including Biofeedback, Osteopathic Procedures, Behavioral Training, Diet Control, and Electrical Stimulation in the Management of Urinary Incontinence in Children With Lumbar or Sacral Myelomeningocele Spina Bifida: A Randomized Controlled Trial
Brief Title: Effectiveness of Multimodal Therapy for Urinary Incontinence in Pediatric Spina Bifida
Acronym: MMICIUISP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hany Mohamed Ibrahim Elgohary, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00014233-56
Record Dates: First submitted 2026-01-04; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Myelomeningocele Spina Bifida
Keywords: Urinary Incontinence; Pelvic Floor; Electromyography; Quality of Life; Child
MeSH Terms: conditions — Urinary Incontinence | interventions — Diet; Electric Stimulation Therapy

STUDY DESIGN:
Intervention Model Description: Study Design The current study was designed as a randomized, controlled, parallel-group clinical trial between May 2024 and August 2025. The definitive aim of the study was to evaluate the efficacy of a multimodal rehabilitation program-biofeedback training, osteopathic treatment, behavioral modification, dietary control, and interferential current therapy-in urinary incontinence of pediatric patients with lumbar or sacral myelomeningocele spina bifida. The participants were randomly assigned using a computer-generated randomization list of two equal groups of participants. Group A was exposed to the multimodal intervention and group B to the conventional physiotherapeutic intervention based on the pelvic-floor muscle training and educative program. The concealment of allocation was carefully maintained by use of sequentially numbered, opaque and sealed envelopes which were under the care of an independent researcher who did not take part in the process of data acquisition and data
Masking Description: Blinding was preserved to the level of outcome assessors and statisticians who were not aware of the group assignments during the intervention and the analytical stage.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): 1. Diet and Toileting Education The implementation of the intervention was based on behavioral interventions, including diet and toileting education. In the first session, both children and their caregivers were provided with personalized counseling on the need to balance the intake of fluids and dietary fiber within the age specifications. The guidelines recommended that people always should take fruits, vegetables, and whole grains and avoid constipating foods like high dairy and refined carbohydrates. children were taught to promote regular toileting routines especially planned toileting which lasts about ten minutes after meals with foot support to enhance the pelvis positioning and defecation dynamics. Reward chart system was implemented to strengthen the adherence and promote good toileting behaviors. This was followed by weekly reinforcement sessions before to check the progress, dietary questions and modify recommendations. Adherence was monitored by using caregiver diaries
  Interventions: Other: Diet and Toileting Education; Other: Pelvic Floor Physiotherapy; Other: Abdominal Strengthening Program.; Other: Interferential Current Therapy; Other: Osteopathy Protocol; Other: Biofeedback Training Procedure.
- Group B (Active Comparator): Pelvic Floor Physiotherapy Certified pediatric physiotherapists administered pelvic floor muscle (PFM) physiotherapy, twice a week, during 8 weeks. Every session started with an education on the anatomy and physiology of the bladder and pelvic floor with focus on the normal voiding patterns and how relaxation and contraction are used to manage continence. The first sessions aimed at down-training the maladaptive voiding postures with visual and tangible feedback to correct the maladaptive posture and enhance awareness. Environmental training was active training that comprised of blow-out-candle breathing exercises to coordinate the abdominal push with pelvic-floor relaxation by three sets of 8 -12 reps which were practiced both morning and evening at home. Surface EMG biofeedback was used, in 8 sessions of supervision to give a visual representation of muscle control and involvement. The participants were advised to keep exercise records and were given parental coaching
  Interventions: Other: Diet and Toileting Education; Other: Pelvic Floor Physiotherapy

INTERVENTIONS:
Other: Diet and Toileting Education — The implementation of the intervention was based on behavioral interventions, including diet and toileting education. In the first session, both children and their caregivers were provided with personalized counseling on the need to balance the intake of fluids and dietary fiber within the age specifications. The guidelines recommended that people always should take fruits, vegetables, and whole grains and avoid constipating foods like high dairy and refined carbohydrates. children were taught to promote regular toileting routines especially planned toileting which lasts about ten minutes after meals with foot support to enhance the pelvis positioning and defecation dynamics. Reward chart system was implemented to strengthen the adherence and promote good toileting behaviors. This was followed by weekly reinforcement sessions before to check the progress, dietary questions and modify recommendations. Adherence was monitored by using caregiver diaries and or
Other: Pelvic Floor Physiotherapy — Certified pediatric physiotherapists administered pelvic floor muscle (PFM) physiotherapy, twice a week, during 8 weeks. Every session started with an education on the anatomy and physiology of the bladder and pelvic floor with focus on the normal voiding patterns and how relaxation and contraction are used to manage continence. The first sessions aimed at down-training the maladaptive voiding postures with visual and tangible feedback to correct the maladaptive posture and enhance awareness. Environmental training was active training that comprised of blow-out-candle breathing exercises to coordinate the abdominal push with pelvic-floor relaxation by three sets of 8 -12 reps which were practiced both morning and evening at home. Surface EMG biofeedback was used, in 8 sessions of supervision to give a visual representation of muscle control and involvement. The participants were advised to keep exercise records and were given parental coaching so that they were practicing at home. Adhe
Other: Abdominal Strengthening Program. — The core and abdominal strengthening program were integrated into physiotherapy programs in a systematic manner. Individualized exercises were based on the motor ability of each child and included the diaphragmatic breathing, gentle isometric abdominal holds (modified dead-bug or bird-dog positions), and seated trunk forward-lean exercises with controlled bear-down maneuvers that were done only with relaxation of the pelvic-floor. Sessions were performed twice a week in the first month and then advanced to a daily 10- 15 minutes. This gradual training was done to improve intra-abdominal pressure management, posture and coordination of respiratory and pelvic muscles to facilitate bladder emptying and continence. The compliance was good and the adherence was documented every week. This aspect supplemented pelvic physiotherapy in restoring neuromuscular coordination and trunk stability that are important in continence mechanisms.
  Arms: Group A
Other: Interferential Current Therapy — IFC sessions were implemented 3 times per week during 8 successive weeks. The duration of every session was 20-30 minutes and used four electrodes; two on the front side of the abdomen above the suprapubic area and two on the back side near the sacral or pelvic-floor area. The frequency used was about 10 kHz to make the interferential waveform more comfortable and acceptable to the patient. The intensity was adjusted to produce a slight tingling feeling without pain and skin integrity was checked on a regular basis. The neuromodulatory effects on detrusor overactivity and sphincter coordination were often combined with pelvic-floor exercises in the same session to enhance the intensity of the neuromodulatory response of IFC.
  Arms: Group A
Other: Osteopathy Protocol — The osteopathic intervention in this study aimed to improve the pelvic position, regain the visceral mobility and the neuromuscular activity in children with lumbar or sacral myelomeningocele-related urinary incontinence. Myofascial, visceral, and articular techniques were included in the osteopathic procedures and each targeted a particular dysfunction in the pelvic and lumbosacral areas. In every 30-minute session, treatments were separated into three combined phases: (1) Myofascial release which involved gentle stretching and inhibition of the psoas muscle and deep-tissue mobilization around the obturator foramen to reduce tension and maximize the movement of the pelvic organs (2) Visceral techniques, including soft-tissue mobilization and stretching of the greater omentum and abdominal viscera to enhance visceral mobility and release fascial restraints that affect bladder and bowel mechanics and (3) Articular mobilization, where high-velocity, low-amplitude (HVLA) manipulations we
  Arms: Group A
Other: Biofeedback Training Procedure. — Biofeedback training, was used as a fundamental element of therapy to improve voluntary control and co-ordination of the PFMs by children with urinary incontinence due to lumbar or sacral myelomeningocele spina bifida. The intervention was performed through surface electromyographic (EMG) biofeedback (Gymna Uniphy N.V., MYO 200, Bilzen, Belgium) that gave real-time visual and auditory feedback of muscle activity. Two cutaneous EMG electrodes were placed at 3 o'clock and 9 o'clock just in front of the anus, which enabled close attention to the contraction patterns of pubococcygeus, iliococcygeus, coccygeus and puborectalis muscles and synergistic activity of the hip flexors, extensors, abdominals, and thigh muscles. A total of 15 minutes for each session was taken, three times a week and in total, 10 weeks were undertaken with a trained pediatric physiotherapist.
  Arms: Group A

SUMMARY:
Background: Overactive bladder and urinary incontinence in children have significant influence on psychosocial well-being and quality of life. The current study compared the effectiveness of the Multimodal Intervention (MMI) protocol to a Conventional Intervention (CI) in increasing urinary control, pelvic floor functioning, and quality of life. 66 adolescents (10-17 years old) were randomly divided into MMI (n=33) and CI (n=33) groups according to the inclusion criteria related to urinary incontinence. A 10-week therapeutic regime was given to every group with a 12-week post-treatment follow-up period. The key outcome measures were the number of urinary incontinence episodes per day, pelvic floor muscle electromyography (EMG) values, voiding frequency, Pediatric Quality of Life Inventory (PedsQL) items, and Pediatric Incontinence Questionnaire (PINQ) items.

DETAILED DESCRIPTION:
Study Design The current study was designed as a randomized, controlled, parallel-group clinical trial between May 2024 and August 2025. The definitive aim of the study was to evaluate the efficacy of a multimodal rehabilitation program; biofeedback training, osteopathic treatment, behavioral modification, dietary control, and interferential current therapy, in urinary incontinence of pediatric patients with lumbar or sacral myelomeningocele spina bifida. The participants were randomly assigned using a computer-generated randomization list of two equal groups of participants. Group A was exposed to the multimodal intervention and group B to the conventional physiotherapeutic intervention based on the pelvic-floor muscle training and educative program. The concealment of allocation was carefully maintained by use of sequentially numbered, opaque and sealed envelopes which were under the care of an independent researcher who did not take part in the process of data acquisition and data analysis.

The study was conducted in the same strict spirit as the principles of ethics as outlined in the Declaration of Helsinki and the institutional ethics committee gave its consent to the research. Written informed consent was presented to parents or legal guardians before the enrolment, and verbal consent was elicited among the children themselves. Blinding was preserved to the level of outcome assessors and statisticians who were not aware of the group assignments during the intervention and the analytical stage.

All participants were thoroughly assessed at the baseline before the intervention and then at the end of the 10-week programmed and 12 weeks later assessed as a follow up. The main outcome measure was the improvement of urinary continuance, measured by the number of the incontinence incidences and thorough analysis of the bladder diaries. The secondary outcomes included pelvic-floor muscle strength (EMG biofeedback measure), voiding behavior and quality of life, measured using the PINQ and the PedsQL. The intervention sessions were conducted in a limited clinical environment through certified pediatric physiotherapists and osteopathic practitioners. All the data were pseudonymized and analyzed accordingly with proper statistical tests to explain within and between group differences.

ELIGIBILITY:
Inclusion Criteria:

* = children with lower lumbar or sacral myelomeningocele spina bifida,
* urinary incontinence due to neurogenic bladder dysfunction
* the ability to understand and adhere to study procedures
* :intelligence required to be engaged in biofeedback and behavioural training activities

Exclusion Criteria

* thoracic or high lumbar myelomeningocele, and other forms of spina bifida with complete sacral loss of innervation
* severe cognitive or behavioral impairments likely to interfere with adherence to training regimens
* uncontrolled epilepsy and severe musculoskeletal deformities that could not allow the placement of the electrode or postural exercises.
* The participants that had undergone urological or neurosurgical operation in the past six months and those who were undergoing botulinum toxin injection or sacral neuromodulation therapy were also disqualified

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 66 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Urinary Continence Improvement | The baseline, post-intervention (week 10), and follow-up (week 12)
  The main outcome of this study was the improvement of urinary continence which was measured by counting the episodes of incontinence recorded in a three-day urinary bladder diary that used a standardized form. The bladder diary is a validated and proven tool of measuring the frequency of urination, voided volumes, and incontinence occurrences in children's studies (Neveus et al., 2019; Austin et al., 2014). It provides objective and subjective information on bladder habits and therapeutic responsiveness. The parents and their children were advised to closely note the wetting and voiding incidences and any accompanying urgency symptoms during three consecutive days before baseline measurement, at the end of the ten-week intervention and at a twelve-week follow-up. The reduction of incontinence rates at the end of the treatment compared to the baseline was directly evaluated as a measure of the effectiveness of treatment and subsequent increase in the quality of bladder control.

SECONDARY OUTCOMES:
Quality of Life (PedsQL) | at the baseline, immediately after the 10 weeks intervention and at 12 weeks follow up
  The influence of urinary incontinence on the child daily functioning and psychosocial well-being was investigated using validated measure, that is PedsQL 4.0, a popular psychometrically sound instrument of health-related quality of life (HRQOL) with internal consistency coefficients of 0.78 to 0.92 within domains (Varni et al., 2001; Eiser and Morse, 2001). The questionnaire was to be conducted at the baseline, immediately after the 10 weeks intervention and at 12 weeks follow up to measure the change in emotional well-being, self-esteem and social participation that might have explained as a result of the therapeutic program.
Pelvic Floor Muscle Strength (EMG Biofeedback) | at the baseline, immediately after the 10 weeks intervention and at 12 weeks follow up
  Pelvic floor muscle (PFM) strength was evaluated using the surface electromyography (EMG) biofeedback through the Gymna Uniphy MYO 200 device (Gymna Uniphy N.V., Bilzen, Belgium). Surface EMG biofeedback is an effective non-invasive, valid, and reliable measure of the neuromuscular activity of the pelvic floor and associated musculature of pediatric populations (Bo and Sherburn 2005; Glazer, 1999). To record voluntary contractions and relaxation of the pelvic floor muscles as the child followed visual and auditory signals, two electrodes as adhesive surfaces were placed perianal at the 3- and 9-hour positions. PFM strength was measured using the peak amplitude (µV) and contraction duration. The baseline, post-intervention (week 10), and follow-up (week 12) were measured to assess the progression and the maintenance of the neuromuscular improvements.

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of physical therapy, Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
It will be available when needed

REFERENCES:
- See also: Related Info — https://orcid.org/0000-0001-5531-1875